CLINICAL TRIAL: NCT03293056
Title: Effectiveness of High-intensity Interval Versus Intensity Continuous Hydrogymnastics for Improvement of Health Outcomes: Randomized Clinical Trial.
Brief Title: HIIH Versus HMC: Randomized Clinical Trial
Acronym: HIITxHMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do vale do São Francisco (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Rodrigo Gustavo da Silva Carvalho, Rodrigo Gustavo da Silva Carvalho, Universidade Federal do vale do São Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012017
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Healthy People
Keywords: aerobic exercises; training; aquatic

STUDY DESIGN:
Intervention Model Description: Parallel Assignment: highintensity interval training water versus aerobic continuous
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity Interval Hydrogynmastics (Experimental): High-intensity Interval training Hydrogynmastics, 2x/week, for 3 months.
  Interventions: Other: High-intensity interval Hydrogynmastics
- Hydrogynmastics Continuous Moderate (Active Comparator): Hydrogynmastics Continuous Moderate training (HCM), 2x/week, for 3 months.
  Interventions: Other: Hydrogynmastics Continuous Moderate

INTERVENTIONS:
Other: High-intensity interval Hydrogynmastics — The HIIH to PSE group during the high intensity (HI) period should remain between 16 to 18 points, while in the moderate intensity (MI) intervals around 11. The dynamic exercises will progression, in the first month will be 1 min of HI and 2 min of MI, in the second month of 1 min of HI and 1 min of MI and in the last month of 1 min of HI and 30 s of MI, until completing 30 min in total.
  Other Names: HIIH
  Arms: High-intensity Interval Hydrogynmastics
Other: Hydrogynmastics Continuous Moderate — For the HCM group the PSE will be around 11 points during the 30 min of moderate continuous exercise. In both groups the form of intensity monitoring that will be through the PSE, in which this scale will be printed in banner form and affixed next to the physical education teacher during the classes.
  Other Names: HCM
  Arms: Hydrogynmastics Continuous Moderate

SUMMARY:
Introduction: water aerobics involves the practice of specific aquatic exercises that are based on the use of water resistance as a load and on thrust as an impact reducer, making it possible to perform physical exercise with a lower risk of injury even at a high intensity. Objective: The overall objective of this study will be to compare the effectiveness of high intensity interval versus moderate continuous water aerobics to improve health outcomes in apparently healthy individuals.

DETAILED DESCRIPTION:
Method: randomized clinical trial will be performed in the premises of the College of Physical Education of the Federal University of the São Francisco Valley. 100 adults, of both sexes, will be randomized into two groups, high intensity interval hydrogynastic (HIAI) or moderate continuous aquatic gymnastics (HCM). Individuals will be evaluated for primary endpoints of muscle strength and endurance, aerobic fitness, flexibility and body composition. The secondary outcomes evaluated will be the quality of life, functionality and perception of improvement by a Likert-type Improvement Scale, at the following moments: initial, final and follow-up of one month after the end of the training. Individuals will be assisted for three months, often weekly twice, with sessions lasting 50 min. In order to identify differences between and within the groups, an equation of generalized estimates will be used as regression model with the syntax according to the multivariate model.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60 years;
* sedentary and who did not perform physiotherapy and physical activity in the last three months;
* clinical and cognitive conditions for swimming pool activities and aerobic exercise; who have not undergone highly complex surgical procedures in the last six months;
* to be able of walking without help equipment and without musculoskeletal or skeletal diseases;
* without contraindications to the practice of exercises; such as: urinary and / or fecal incontinence and dermatological diseases;
* below obesity II with BMI <40.

Exclusion Criteria:

* if they have up to three consecutive fouls during the hydrogymnastics period;
* if they present any adverse effects, such as: allergy or any dermatitis;
* unable to continue the study due to change of address or hospitalization.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Aerobic Fitness | three months after randomization
  This maximal/submaximal test will be performed on cyclergometer, Balke test.
Body Composition | three months after randomization
  The body composition (density and percentage of body fat) will be estimated by prediction equations (JACKSON et al., 1980).
Strength Muscular | three months after randomization
  Strength Muscular will be measured by 1RM test in two exercises, involving the segments of the upper limbs (supine) and lower limbs (leg press).
Endurance Muscular | three months after randomization
  Muscle endurance will be assessed by the test in which the individual performs the maximum number of repetitions of given exercises for one minute. The exercises will be of arm and abdominal flexion.

SECONDARY OUTCOMES:
Quality Life | three months after randomization
  Quality of life by assessed by WHOQOL-breaf
Functionality | three months after randomization
  Functionality will be assessed by IVCF-20
Perception of Improvement | three months after randomization
  Perception of Improvement will be measured by an Likert-type Improvement Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Education College, Petrolina, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No